CLINICAL TRIAL: NCT06819969
Title: The Canadian Lung Outcomes in Users of Vaping Devices (CLOUD) Study
Brief Title: The Canadian Lung Outcomes in Users of Vaping Devices Study
Acronym: CLOUD
Status: Not yet recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: BC Children's Hospital Research Institute (Other); Providence Healthcare (Other); British Columbia Cancer Agency (Other); University of Alberta (Other); McMaster University (Other); University of Ottawa (Other); Université de Sherbrooke (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Janice Leung, Assistant Professor, Department of Medicine, University of British Columbia, Principal Investigator, Centre for Heart Lung Innovation, St. Paul's Hospital, Respirologist, St. Paul's Hospital, University of British Columbia
Other Study IDs: H24-00374; FRN-193735 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR)); FRN-193735 (Other Grant/Funding Number: Heart and Stroke Foundation); FRN-193735 (Other Grant/Funding Number: Canadian Cancer Society)
Record Dates: First submitted 2025-01-27; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Small Airways Diseases; Vaping; Vaping Related Disorder; Vaping Teens; Vaping Behavior
Keywords: CLOUD; small airway injury; vaping; vape; e-cigarette; oscillometry; multiple breath washout; chest computed tomography; chest CT; hyperpolarized 129-xenon; MRI; CPET; bronchoscopy; transcriptomics; epigenetics
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All cohorts: Blood Adolescent cohort: Induced Sputum Adult cohort: Airway Epithelium and Lung Immune Cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adults: Canadian adults aged 19 years or older. We will be enrolling e-cigarette-only users, non-e-cigarette and non-combustible cigarette users, combustible cigarette-only users, and dual combustible cigarette-e-cigarette users.
- Adolescents: Canadian adolescents aged between 12 and <19 years, inclusive. We will be enrolling e-cigarette-only users, as well as non-e-cigarette and non-combustible cigarette users.

SUMMARY:
Vaping is increasingly popular with both adolescent and adult Canadians, but the long-term health impacts remain unknown. We believe that the tools we currently have to detect lung disease in people who vape may be insufficient and propose new ways to find lung injuries that may impact them over the course of their lives. These include exercise testing, new imaging techniques, and new breathing tests that will demonstrate how vaping may harm their lungs. We will use these tools in both adolescent and adult Canadians to give Canadians who vape important information on the consequences of vaping.

DETAILED DESCRIPTION:
Promoted as a safer method of inhaling nicotine compared to cigarettes and as smoking cessation tools, e-cigarettes have substantially grown in popularity with rates of uptake now exceeding those of cigarette smoking. In Canada, 6% of Canadians aged 15 years and older have vaped in the past 30 days. Younger Canadians appear to be the most susceptible to these habits, with 14% of those aged 15-19 years and 18% of those aged 20-24 years reporting past 30 day use. Indigenous populations are also disproportionately affected by the spread of vaping which may place them at higher risk for potential downstream respiratory complications. As Canadians increasingly reach for e-cigarettes, especially at younger ages and not just for the purposes of smoking cessation, greater clarity into the pulmonary toxicities vaping is urgently needed.

The Canadian Lung Outcomes in Users of Vaping Devices (CLOUD) Study is a pan-Canadian, multicentre, multidisciplinary, and longitudinal approach to studying vaping from cell to society. The characterization of e-cigarettes' respiratory effects remains superficial and a more comprehensive phenotyping of vaping-exposed lungs across the lifespan using novel imaging and pulmonary function techniques, dynamic exercise testing, and airway cell sequencing would significantly enhance our understanding of the potential harms. As with combustible cigarette smoking, the small airways (characterized by a diameter <2mm) may be particularly vulnerable during vaping given their high degree of exposure to particulate matter. These regions of the lung may harbour the earliest signs of injury, ultimately setting the stage for future obstructive airways disease.

Objectives

The objective of the CLOUD Study is to characterize small airway injury in adolescent and adult Canadians who use e-cigarettes. Specifically, our goals are to:

1. Characterize the structural and functional disruptions associated with e-cigarette use using oscillometry, multiple breath washout, chest computed tomography, hyperpolarized 129-xenon magnetic resonance imaging, cardiopulmonary exercise testing, and bronchoscopy.
2. Determine the association between e-cigarette use and respiratory outcomes, including symptom burdens, exacerbation-like respiratory events, and school and work absences.
3. Characterize the epigenetic and transcriptomic disruptions associated with e-cigarette use in blood, sputum, airway epithelium, and lung immune cells.

Methods Our observational, longitudinal cohort study encompasses six academic hospital centres across Canada (the University of British Columbia, the University of Alberta, McMaster University, the University of Ottawa, the University of Toronto, and the Université de Sherbrooke). Participants (n=100 ages >12 and <19 years and n=400 ages ≥19 years) will be followed over 3 years, undergoing repeat demographic and respiratory symptom questionnaires, oscillometry, pulmonary function testing, and exercise testing. Adolescent participants will additionally undergo multiple breath washout and induced sputum collection and adult participants will undergo chest CT imaging and bronchoscopy. A substudy of adolescent and adult participants undergoing pulmonary hyperpolarized 129-xenon gas magnetic resonance imaging will also be performed. Induced sputum and bronchoscopy-derived airway epithelial and bronchoalveolar lavage samples will be sequenced for methylation and transcriptomics.

ELIGIBILITY:
Inclusion Criteria:

Adolescent arm:

* Aged ≥12 and <19 years old
* Either 1) use neither combustible cigarettes nor e-cigarettes or 2) use e-cigarettes exclusively

Adult arm:

* Aged ≥19 years old
* Fall into one of the following categories: 1) use neither combustible cigarettes nor e-cigarettes; 2) use combustible cigarettes exclusively, never using e-cigarettes; 3) use e-cigarettes exclusively, never using combustible cigarettes; or 4) use both combustible cigarettes and e-cigarettes currently

Exclusion Criteria:

Adolescent arm:

* Contraindication to pulmonary function testing and cardiopulmonary exercise testing
* Have smoked combustible cannabis within the last month and/or have a combustible cannabis smoking history of >1 joint-year
* Have smoked combustible cigarettes within the last 6 months
* Have a physician-diagnosed chronic lung disease (such as asthma, cystic fibrosis, or bronchopulmonary dysplasia)
* Inability to provide written informed consent

Adult arm:

* Contraindication to pulmonary function testing and cardiopulmonary exercise testing
* Have smoked combustible cannabis within the last month and/or have a combustible cannabis smoking history of >1 joint-year
* Currently undergoing treatment for lung cancer
* Inability to provide written informed consent

No limitations will be placed on the type of e-liquids used by participants; e.g., e-cigarette users of nicotine, tetrahydrocannabinol, and cannabidiol will be all enrolled.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll both adolescent (ages ≥12 and <19 years) and adult (≥19 years) e-cigarette and non-e-cigarette users in six academic hospital centres across Canada.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Composite Measure of Small Airways Dysfunction | From enrollment (Baseline) to the end of study participation (36 Months).
  Participants meeting at least one of the following criteria will be considered to have small airways dysfunction:
  For adolescent participants, these measures will include 1) a change in resistance from 5-20 Hz (R5-R20) >upper limit of normal (ULN) on oscillometry or 2) peak oxygen consumption (VO2)<lower limit of normal (LLN) plus a ventilatory response or minute ventilation/carbon dioxide production (VE/VCO2) nadir >ULN. For adult participants, these measures will include 1) R5-R20 >ULN, 2) disease probability measure functional small airways disease >10% on chest CT, or 3) peak VO2<84% predicted plus a VE/VCO2 nadir >ULN. The proportion of participants meeting at least one of the criteria for small airways dysfunction at any time point will be compared between the vaping and control groups using Chi-square tests. Multivariable logistic regressions will be used to adjust for possible covariates, such as age, sex, and their interaction with vaping/smoking groups.

SECONDARY OUTCOMES:
FEV1 | 36 Months
  Outcome measured in units of Liters (L) for all study participants.
FVC | 36 Months
  Outcome measured in units of Liters (L) for all study participants.
FEV1/FVC | 36 Months
  Outcome measured in units of 0-100% for all study participants.
FEV3/FEV6 | 36 Months
  Outcome measured in units of 0-100% for all study participants.
Total Lung Capacity | 36 Months
  Outcome measured in units of Liters (L) for all study participants.
Diffusion Capacity | 36 Months
  Outcome measured in units of mL/min/mmHg for all study participants.
Small Airways Resistance R5-R20 | 36 Months
  Outcome measured in units of kPa/l/s for all study participants.
Ventilation Defect Percent | 36 Months
  Outcomes measured in units of 0-100% for study participants in the following sites: St. Paul's Hospital (University of British Columbia), BC Children's Hospital (University of British Columbia), the Hospital for Sick Children (University of Toronto), St. Joseph's Healthcare Hamilton (McMaster University).
RBC to Membrane Ratio | 36 Months
  Outcomes measured in units of a ratio for study participants in the following sites: St. Paul's Hospital (University of British Columbia), BC Children's Hospital (University of British Columbia), the Hospital for Sick Children (University of Toronto), St. Joseph's Healthcare Hamilton (McMaster University).
Membrane to Gas Ratio | 36 Months
  Outcomes measured in units of a ratio for study participants in the following sites: St. Paul's Hospital (University of British Columbia), BC Children's Hospital (University of British Columbia), the Hospital for Sick Children (University of Toronto), St. Joseph's Healthcare Hamilton (McMaster University).
Apparent Diffusion Coefficient | 36 Months
  Outcomes measured in units of cm2/s for study participants in the following sites: St. Paul's Hospital (University of British Columbia), BC Children's Hospital (University of British Columbia), the Hospital for Sick Children (University of Toronto), St. Joseph's Healthcare Hamilton (McMaster University).
Peak VO2 %predicted | 36 Months
  Outcomes measured in units of 0-100% for all study participants.
VE/VCO2 nadir | 36 Months
  Outcomes measured in units of a ratio for all study participants.
Epigenetic Age (Blood Methylation) | 36 Months
  Outcomes measured in units of age acceleration residual for all study participants.
Differentially Methylated Genes (Blood Methylation) | 36 Months
  Outcomes measured in units of beta-values for all study participants.
Differentially Expressed Genes (Blood Transcriptome) | 36 Months
  Outcomes measured in units of transcripts per million for all study participants.
Epigenetic Age (Induced Sputum Methylation) | 36 Months
  Outcomes measured in units of age acceleration residual for adolescent study participants in the following sites: BC Children's Hospital (University of British Columbia), the Hospital for Sick Children (University of Toronto), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke).
Differentially Methylated Genes (Induced Sputum Methylation) | 36 Months
  Outcomes measured in units of beta-values for adolescent study participants in the following sites: BC Children's Hospital (University of British Columbia), the Hospital for Sick Children (University of Toronto), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke).
Differentially Expressed Genes (Induced Sputum Transcriptome) | 36 Months
  Outcomes measured in units of transcripts per million for adolescent study participants in the following sites: BC Children's Hospital (University of British Columbia), the Hospital for Sick Children (University of Toronto), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke).
Epigenetic Age (Bronchial Epithelial Cell and Bronchoalveolar Lavage Methylation) | 36 Months
  Outcomes measured in units of age acceleration residual for adult study participants in the following sites: St. Paul's Hospital (University of British Columbia), St. Joseph's Healthcare Hamilton (McMaster University), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke).
Differentially Methylated Genes (Bronchial Epithelial Cell and Bronchoalveolar Lavage Methylation) | 36 Months
  Outcomes measured in units of beta-values for adult study participants in the following sites: St. Paul's Hospital (University of British Columbia), St. Joseph's Healthcare Hamilton (McMaster University), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke).
Differentially Expressed Genes (Bronchial Epithelial Cell and Bronchoalveolar Lavage Transcriptome) | 36 Months
  Outcomes measured in units of transcripts per million for adult study participants in the following sites: St. Paul's Hospital (University of British Columbia), St. Joseph's Healthcare Hamilton (McMaster University), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke).
Lung Clearance Index | 36 Months
  Outcomes measured in counts for adolescent study participants in the following sites: BC Children's Hospital (University of British Columbia), the Hospital for Sick Children (University of Toronto).
DPM fSAD | 36 Months
  Outcomes measured in units of 0-100% for adult study participants in the following sites: St. Paul's Hospital (University of British Columbia), St. Joseph's Healthcare Hamilton (McMaster University), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke), Clinical Sciences Building (University of Alberta), Ottawa Hospital General Campus (University of Ottawa).
LAA856 | 36 Months
  Outcomes measured in units of 0-100% for adult study participants in the following sites: St. Paul's Hospital (University of British Columbia), St. Joseph's Healthcare Hamilton (McMaster University), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke), Clinical Sciences Building (University of Alberta), Ottawa Hospital General Campus (University of Ottawa).
LAA950 (Quantitative Emphysema) | 36 Months
  Outcomes measured in units of 0-100% for adult study participants in the following sites: St. Paul's Hospital (University of British Columbia), St. Joseph's Healthcare Hamilton (McMaster University), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke), Clinical Sciences Building (University of Alberta), Ottawa Hospital General Campus (University of Ottawa).
Qualitative Emphysema | 36 Months
  Outcomes measured in units of 0-100% for adult study participants in the following sites: St. Paul's Hospital (University of British Columbia), St. Joseph's Healthcare Hamilton (McMaster University), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke), Clinical Sciences Building (University of Alberta), Ottawa Hospital General Campus (University of Ottawa).
Pulmonary Vascular Volume | 36 Months
  Outcomes measured in units of milliliters (mL) for adult study participants in the following sites: St. Paul's Hospital (University of British Columbia), St. Joseph's Healthcare Hamilton (McMaster University), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke), Clinical Sciences Building (University of Alberta), Ottawa Hospital General Campus (University of Ottawa).
Mucus Score | 36 Months
  Outcomes measured in counts for adult study participants in the following sites: St. Paul's Hospital (University of British Columbia), St. Joseph's Healthcare Hamilton (McMaster University), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke), Clinical Sciences Building (University of Alberta), Ottawa Hospital General Campus (University of Ottawa).
Total Airway Counts | 36 Months
  Outcomes measured in counts for adult study participants in the following sites: St. Paul's Hospital (University of British Columbia), St. Joseph's Healthcare Hamilton (McMaster University), Centre Hospitalier Universitaire de Sherbrooke (Universite de Sherbrooke), Clinical Sciences Building (University of Alberta), Ottawa Hospital General Campus (University of Ottawa).

CONTACTS AND LOCATIONS:
Overall Officials: Janice Leung, MD, Principal Investigator — University of British Columbia
Locations (8):
- Canada (8):
  - University of Alberta (Clinical Sciences Building), Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - BC Children's Hospital Research Institute, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - McMaster University (Research Institute of St. Joe's Hamilton), Hamilton, Ontario
  - University of Ottawa (The Ottawa Hospital General Campus), Ottawa, Ontario
  - University of Toronto (The Hospital for Sick Children), Toronto, Ontario
  - Université de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burns P, Eddy RL, Li X, Yang J, Dhillon SS, Couillard S, Stickland MK, Guenette J, Svenningsen S, Tulloch T, Samji H, Meza R, Struik LL, Aaron S, Ho T, Lam S, Leipsic J, Maclean J, Afshar T, Moraes TJ, Zanette B, Santyr G, Counil FP, Hernandez Cordero AI, Matano S, de Arruda Maluf G, Leung C, Feng C, Bal L, Dhaliwal H, Mumuni A, Lui C, Drew H, Sin DD, Rayment JH, Leung JM. The Canadian Lung Outcomes in Users of Vaping Devices (CLOUD) Study: protocol for a prospective, observational cohort study. BMJ Open. 2025 Mar 6;15(3):e100568. doi: 10.1136/bmjopen-2025-100568. PMID 40050062
- See also: CLOUD Study website containing all details and contact information related to the study. — https://www.cloudstudy.ca/